CLINICAL TRIAL: NCT06156553
Title: School-based Intervention to Support Active Travel. This Study is Part of the Research Project "ULSE - Promoting Active School Travel to Improve Mood and Performance".
Brief Title: School-based Intervention to Support Active Travel
Acronym: PULSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Institute for Studies of Innovation, Research and Education (Other)
Collaborators: The Institute of Transport Economics, Norway (Unknown); University of Agder (Other); Fredrikstad municipality, Norway (Unknown); INSPIRIA Science Center, Norway (Unknown)
Responsible Party: Principal Investigator, Cathrine Pedersen, Senior researcher, Nordic Institute for Studies of Innovation, Research and Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21364
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Physical Inactivity; Health Literacy
Keywords: Active travel; Curriculum-based school intervention; Feasibility study
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Students in 9. grade participating in a school-based intervention (Experimental): Students from 9. grade at 4 schools in a Norwegian municipality. The students will take part in a school and curriculum based intervention delivered by a combination of educators from a science center (1 session) and teachers (5 sessions)
  Interventions: Behavioral: PULSE school-based intervention

INTERVENTIONS:
Behavioral: PULSE school-based intervention — "PULSE - School-based intervention" is a feasibility study designed to support active travel among adolescents. The curricular intervention is designed to increase the students' health literacy as well as their autonomous motivation for active travel. The intervention will last for 6 weeks during fall 2023. The first session will be delivered by a science and education center, and the consecutive sessions will be delivered by teachers. PULSE sessions will contribute to the attainment of specific competence aims related to two interdisciplinary topics, "Health and life skills" and "Sustainability", as defined in PE, social science, and science. The research question is the following: Can increased attention to the barriers and benefits of active travel increase physical activity for youths?

SUMMARY:
"PULSE - School-based intervention" is a feasibility study designed to support active travel among adolescents. The curricular intervention is designed to increase the students' health literacy as well as their autonomous motivation for active travel. The intervention will last for 6 weeks during fall 2023. The first session will be delivered by a science and education center, and the consecutive sessions will be delivered by teachers. PULSE sessions will contribute to the attainment of specific competence aims related to two interdisciplinary topics, "Health and life skills" and "Sustainability", as defined in PE, social science, and science. The research question is the following: Can increased attention to the barriers and benefits of active travel increase physical activity for youths?

DETAILED DESCRIPTION:
Previous reviews and meta-analyses of school-based active travel interventions have found educational strategies to be the most effective. However, previous intervention studies are heterogeneous, and the majority demonstrate poor intervention quality and a lack of description of the interventions. The present study has developed a theory-based educational intervention designed to increase knowledge and empower behavioral change. To ensure local relevance, quality, effectiveness, and sustainability, the intervention has been developed by means of a co-creation process during five collaborative workshops. Participants were a combination of researchers, educators from the science center, representative of the municipality initiative Global Active City in addition to representatives of the teachers from the schools which are to implement the intervention. The intervention is designed to support learning, self-regulation, and autonomous motivation for sustained behavioral change. The theoretical framework is guided by the Self-determination theory developed by Deci and Ryan. The learning activities are predominantly student active and often group-based, introduced by short videos and teacher instructions. The intervention is designed to support three basic psychological needs that, according to the Self-determination theory, are pivotal for motivation and behavioral change: (1) students' need for autonomy and agency related to active travel, (2) their need for relatedness and social support in their efforts to make lifestyle changes when faced with personal, social, and structural barriers, and (3) their need for mastery and competence.

The following data will be collected:

* Questionnaire to students, pre and post
* Document of implementation and adoption completed by teachers
* Group interviews with students who participate in the intervention
* Interviews with teachers who deliver the interviews

ELIGIBILITY:
Inclusion Criteria:

* Student in 9. grade at the 4 intervention schools

Exclusion Criteria:

-

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Active travel habits | 8-10 weeks
  Number of days per week where students walk or use bicycle to/from school or during leisure time activities

SECONDARY OUTCOMES:
Health literacy | 8-10 weeks
  Knowledge about the health benefits of active travel, and where needed information about active travel can be found
Autonomous motivation for active travel | 8-10 weeks
  The students identify with the health, well-being and sustainability benefits of active travel or enjoy their active travels

CONTACTS AND LOCATIONS:
Locations (1):
- NIFU Nordic Institute for Studies of innovation, research and education, Oslo, Norway

REFERENCES:
- See also: Research project website — https://www.nifu.no/prosjekter/pulse-promoting-active-school-travel-to-improve-mood-and-performance/